CLINICAL TRIAL: NCT05289596
Title: Pilot Study: Sleep Well: Implementing an Evidence-Based Digital Insomnia Treatment Program For Physicians
Brief Title: Sleep Well: Digital Insomnia Treatment Program For Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Suzanne M. Bertisch, MD, MPH, Associate Physician and Clinical Director of Behavioral Sleep Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000927
Record Dates: First submitted 2022-02-28; First posted 2022-03-21 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Sleep Disturbance; Insomnia; Stress, Psychological; Anxiety; Burnout, Professional
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; Stress, Psychological; Anxiety Disorders; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evidence-based digital therapy to treat insomnia (Experimental): Participants will be assigned an evidence-based digital therapy to treat insomnia (Sleep Healthy Using the Internet (SHUT-i)
  Interventions: Behavioral: Sleep Healthy Using the Internet (SHUT-i)

INTERVENTIONS:
Behavioral: Sleep Healthy Using the Internet (SHUT-i) — SHUTi is a six session, 6-8 week cognitive behavioral therapy for insomnia program over the internet. The online, self-paced program offers illustrations, graphics, videos and built-in algorithms offering brief sleep diaries, personalized sleep window recommendations, education from sleep experts, peer stories about insomnia, and skills to help participants relearn proper sleep dynamics and increase sleep efficiency.

SUMMARY:
Sleep disturbance is risk factor for incident depression and remains a leading concern for physician burnout; as sleep plays a fundamental role in mood, stress, and cognition, including medical errors. The goal of this project is to implement an evidence-based digital therapy to treat insomnia (Sleep Healthy Using the Internet (SHUTi) for physicians to improve both sleep and mental health outcomes. The investigators will evaluate both process and individual-outcome metrics to define success. Individual level outcomes will be assessed pre-program (at start of participation), week 8 (end-program), and week 16 (2-month follow-up). This information will enable us to design larger future implementation initiatives for the healthy sleep program across the hospital, should the pilot be successful.

DETAILED DESCRIPTION:
The goal of this project is to implement an evidence-based digital therapy to treat insomnia (Sleep Healthy Using the Internet (shut-i) for physicians to improve both sleep and mental health outcomes. The investigators will evaluate both process and individual-outcome metrics to define success. This information will enable us to design larger future implementation initiatives for the healthy sleep program across the hospital, should the pilot be successful. The investigators plan to enroll 25 physicians who screen positive for insomnia (ISI >7). Interested potential participants will complete a preliminary screening to assess eligibility. Refusal rates and eligibility status will be tracked for recruitment yields.

Recruitment will be done via hospital newsletters, information boards, emails, and faculty meetings. Screening will be done through self-service digital questionnaire. Eligible participants will review an e-consent factsheet (REDCap).

Those who enroll will complete surveys at baseline (pre-program), week 8 (end of program), and week 16 (2-month follow-up) securely via REDCap. In addition, feasibility and acceptability data based on the RE-AIM framework and a sub-sample of participants will be invited to an optional intervention feedback interview.

The investigators will evaluate the feasibility and acceptability of recruiting from our target population, delivering our intervention with high adherence and fidelity, and estimating effect sizes of our patient-reported outcomes, including sleep duration, quality, mood, and burnout. Assessment criteria will be based on the RE-AIM model for program evaluation (reach, effectiveness, adoption, implementation, maintenance).

It will be the responsibility of the PI to oversee the safety of the study. The PI will follow the Partners' policy Reporting Unanticipated Problems including Adverse Events (Rev. 9/24/2014) and will promptly report problems to the PHRC.

ELIGIBILITY:
Inclusion Criteria:

* Have a digital device with reliable internet access
* Physician within the BWH Physician Organization
* Insomnia Severity Index (ISI) score ≥8
* Able to give informed consent

Exclusion Criteria:

* Shift work >1 day/week over the treatment course
* Excessive daytime sleepiness (ESS≥16)
* History of bipolar disorder
* History of seizure within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance, 8b | 10 weeks
  PROMIS Sleep Disturbance measures self-reported sleep quality and associated daytime functioning during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance. The minimum score is 8 and the maximum score is 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
PROMIS Sleep Impairment, 8a | 10 weeks
  PROMIS Sleep Impairment measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness during the past seven days. The measure includes 8-items with higher scores indicating greater sleep impairment. The minimum score is 8 and the maximum score 40. Item responses are combined to yield a T-score with a population mean of 50 and standard deviation of 10.
Insomnia Severity Index, ISI | 10 weeks
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Bertisch, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Benge E, Lauffenburger JC, Reid M, Rottapel R, Mehta D, Bertisch SM. Leveraging digital therapeutics to improve physician sleep: a pilot implementation study. J Clin Sleep Med. 2025 Jul 1;21(7):1297-1299. doi: 10.5664/jcsm.11666. PMID 40114469